CLINICAL TRIAL: NCT03993678
Title: Intratumoral Injection of IP-001 Following Thermal Ablation in Patients With Advanced Solid Tumors. A Multicenter Phase Ib/IIa Trial With Expansion Cohorts in Melanoma and Soft Tissue Sarcoma Patients.
Brief Title: Intratumoral Injection of IP-001 Following Thermal Ablation in Patients With Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Collaborators: Immunophotonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 66/17
Record Dates: First submitted 2019-06-18; First posted 2019-06-21 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors
Keywords: advanced solid tumors; Intratumoral injection; IP-001; thermal ablation; phase Ib/IIa; melanoma; soft tissue sarcoma; tumor ablation; systemic immune response; interventional immuno-oncology; abscopal effect; T cell stimulation
MeSH Terms: conditions — Melanoma; Sarcoma | interventions — N-dihydrogalactochitosan; Transurethral Resection of Prostate

STUDY DESIGN:
Intervention Model Description: Multicenter single arm, phase Ib/IIa with 2 Parts:
  * Part 1 (referring to the phase Ib part of the trial) consists of a safety run-in cohort with 1 dose level (DL) of IP-001 and a de-escalation safety step with a reduced dose of IP-001, if needed. This 'all-comers' cohort will enroll patients with laser ablation-accessible advanced solid tumors.
  * Part 2
    * Cohort 1: Dose expansion cohort consisting of 9 patients with advanced STS treated at the tentative recommended phase 2 dose (RP2D), as established in Part 1;
    * Cohort 2: Phase IIa part consisting of 18 patients with advanced melanoma treated at the tentative RP2D, as established in Part 1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ablation + IP-001 (Experimental): Ablation + IP-001 will be administered every 4 weeks for up to 6 treatment visits.
  Trial treatment will stop in case of tumor progression according to RECIST 1.1 or iRECIST or unacceptable toxicity.
  In all cases, toxicity assessment will continue for at least 100 days after discontinuing the last treatment of Ablation + IP-001 or until resolution of Ablation + IP-001-associated toxicity.
  Interventions: Drug: IP-001; Device: Thermal Ablation

INTERVENTIONS:
Drug: IP-001 — Dose and route: Immediately (within 15 - 30 min) after thermal ablation, IP-001 will be injected in and around the ablated lesion. The amount of IP-001 injected depends on the dose level.
Device: Thermal Ablation — The medical device includes a laser unit. The system continuously measures the temperature of the tissue, guiding the user to perform precise and safe treatments.
  Treatment time: 30 min
  Other Names: TRANBERG Thermal Therapy System®; Thermal Therapy System (Clinical Laserthermia Systems AB)

SUMMARY:
The therapeutic approach taken by trial SAKK 66/17 is different from those already used in clinical practice and possibly offers patients a therapeutic benefit after failure of standard chemotherapy and immunotherapy.

Patients with laser ablation-accessible solid tumors are treated by thermal ablation followed immediately by an intratumoral injection of IP-001 (1 % N-dihydro-galacto-chitosan, Immunophotonics Inc.) for injection). IP-001 is intended to trigger a tumor-specific systemic immune response when exposed to tumor antigens liberated by thermal ablation. There is strong preclinical and early clinical evidence that combining thermal ablation with IP-001 might be able to turn 'cold' tumors into 'hot' tumors, inducing a systemic immune response. This may result in shrinkage of the treated tumor, as well as, long-term response mediated by the patient's immunological defense system against any remaining tumor cells (residual primary and metastatic tumor cells) including tumor cells outside or distant from the treated area (also known as abscopal effect).

This trial will provide information on the safety and tolerability of thermal ablation followed immediately by an intratumoral IP-001 injection (Ablation + IP-001) in patients with laser ablation-accessible solid tumors ('all comers', Part 1 - safety run in). Further information on safety and tolerability, as well as preliminary antitumor activity, will be evaluated in patients with soft tissue sarcoma (Part 2, Cohort1), whereas in melanoma patients, anti-tumor activity will be defined as a primary objective (Part 2, Cohort 2).

The trial treatment consists of an Ablation + IP-001 in 4-week intervals for up to 6 scheduled treatments. Thermal ablation will be performed according to the instruction of the medical device, and IP-001 will be administered in different dose levels according to the trial design. All patients will be followed until progression of disease or until the start of a subsequent treatment.

DETAILED DESCRIPTION:
Despite constant progress in the treatment of patients with advanced solid tumors failing standard systemic treatment, there is still a high unmet medical need to develop new active anticancer drugs or therapies. Although patients with advanced melanoma have benefitted substantially from the new checkpoint inhibitors, monoclonal antibodies, etc., those patients progressing after such treatment are still in high need of additional treatment options. In the field of advanced sarcoma, little to no progress has been made in the last years, and chemotherapy is still standard treatment for these patients. The therapeutic approach taken by trial SAKK 66/17 is different from those already used in clinical practice and possibly offers patients a therapeutic benefit after failure of standard chemotherapy and immunotherapy. There is strong preclinical and early clinical evidence that combining thermal ablation with IP-001 (1 % N-dihydro-galacto-chitosan, Immunophotonics Inc.) for injection) might be able to turn 'cold' tumors into 'hot' tumors, inducing a systemic immune response. This may result in shrinkage of the treated tumor, as well as long-term response mediated by the patient's immunological defense system against any remaining tumor cells (residual primary and metastatic tumor cells), including tumor cells outside or distant from the treated area (also known as abscopal effect).

The primary objective of Part 1 is to determine the safety and tolerability of thermal ablation followed immediately by an intratumoral IP-001 injection (Ablation + IP-001) in patients with laser ablation-accessible solid tumors ('all comers').

The primary objective of Part 2 - Cohort 1 (soft tissue sarcoma, STS) is to further determine the safety and tolerability of thermal ablation followed immediately by an intratumoral IP-001 injection (Ablation + IP-001) in the dose established in Part 1 of the trial.

The primary objective of Part 2 - Cohort 2 (melanoma) of the trial is to define anti-tumor activity of thermal ablation followed immediately by an intratumoral IP-001 injection (Ablation + IP-001) utilizing the dose established in Part 1 of the trial.

The secondary objective of the trial is

* to further determine the safety and tolerability of IP-001 (Part 2, Cohort 1 and 2)
* to assess the preliminary anti-tumor activity in STS patients (Part 2, Cohort 1)
* to observe further signs of clinical preliminary anti-tumor activity in patients with melanoma (Part 2, Cohort 2).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and ICH/GCP regulations before registration.
* Part 1: - 'All comer' Patients with either histologically or cytologically confirmed advanced or recurrent solid tumor cancer who failed standard therapy, are not eligible for standard therapy, or for whom no effective standard therapy is available and not requiring fast responses.
* Part 2, Cohort 1 - Sarcoma cohort: Patients with either histologically or cytologically confirmed advanced or recurrent soft tissue sarcoma who failed standard therapy, are not eligible for standard therapy or for whom no effective standard therapy is available.
* Part 2, Cohort 2 - Melanoma cohort: Patients with either histologically or cytologically confirmed advanced or recurrent melanoma who failed standard therapy (including a BRAF inhibitor for BRAF-mutant patients), are not eligible for standard therapy or for whom no effective standard therapy is available and have LDH < ULN.
* Presence of at least one tumor lesion that is laser ablation-accessible, with a minimum size of 1.0 cm and located (typically subcutaneously) that it can be treated with Ablation + IP-001 without risk of skin necrosis or serious damage to other adjacent vital and healthy tissue. This tumor lesion may either belong to the skin, lymph nodes, muscles or subcutaneous tissue.
* Measurable or evaluable disease, determined with the most suitable imaging method (CT, PET-CT or MRI), according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* No evidence of CNS progression for at least 4 weeks after completion of CNS-directed therapy as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period.
* Age ≥ 18 years
* WHO performance status 0-2
* Bone marrow function: neutrophil count ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L, hemoglobin ≥ 90 g/L
* Hepatic function: bilirubin ≤ 1.5 x ULN, aspartate transaminase (AST) and alanine transaminase ALT ≤ 2.5 x ULN (or ≤ 5 x ULN in presence of liver metastasis)
* Renal function: estimated glomerular filtration rate (eGFR) > 30 mL/min/1.73m2 (according to Chronic Kidney Disease - Epidemiology Collaboration (CKD-EPI) formula)
* Women with child-bearing potential are using effective contraception, are not pregnant or lactating and agree not to become pregnant during trial treatment and for an additional 90 days after the last dose of investigational drug. Women of childbearing potential must have a negative serum human chorionic gonadotropin (hCG) pregnancy test before inclusion.
* Men agree not to donate sperm or to father a child during trial treatment and until 90 days after the last dose of investigational drug.

Exclusion criteria

* Malignant primary brain tumors, or clinically unstable symptoms from brain metastases or leptomeningeal disease, indicative of active disease.
* Patients who have received chemotherapy, radiotherapy, immunotherapy, or concurrent or recent treatment with any other investigational agents within 21 days (7 days for single fraction of palliative radiotherapy, 42 days for nitrosoureas or mitomycin C) prior to registration.
* Patients who have not recovered to ≤ CTCAE grade 1 from all side effects of prior therapies except for residual toxicities, such as alopecia, which do not pose an ongoing medical risk.
* Patients with a previously treated malignancy, when the risk of the prior malignancy interfering with either safety or efficacy endpoints is not very low.
* Patients with prostate cancer must have discontinued anti-androgens (e.g., bicalutamide, nilutamide) for at least 6 weeks prior to registration; chemical castration with luteinizing hormone-releasing hormone analogues must be continued or patients must be surgically castrated.
* Concomitant treatment with systemic corticosteroids (daily dose of 10 mg prednisolone or equivalent is allowed) or other immunosuppressive therapy (e.g. methotrexate).
* Oral anti-coagulation with vitamin K antagonists (e.g. phenprocoumon, warfarin) and heparin, including therapeutically dosed low molecular weight heparins (LMWH) which cannot be stopped 24 hours prior to trial treatment (low dose aspirin allowed) and bleeding diathesis
* Severe or uncontrolled cardiovascular disease (congestive heart failure New York Heart Association classificationIII or IV), unstable angina pectoris, history of myocardial infarction within the last six months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia), significant QT-prolongation, uncontrolled hypertension .
* Known history of human immunodeficiency virus (HIV) or active chronic Hepatitis C or Hepatitis B Viral infection or any uncontrolled active systemic infection (> CTCAE grade 2) requiring intravenous (iv) antimicrobial treatment
* Serious autoimmune disease (e.g. systemic lupus erythematodes) which is judged to reduce an anti-tumor immune response.
* Known allergic reaction to shellfish, crabs, crustaceans, or any trial components, including medical device, used in trial treatment.
* Any other serious underlying medical, psychological, familial or geographical condition, which in the judgment of the investigator may limit compliance with the planned staging, treatment and follow-up, or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-19 (Actual)

PRIMARY OUTCOMES:
Part 1 and Part 2, cohort 1 (expansion cohort - STS): Dose-limiting toxicity (DLT) | Day 1 to day 28
  The primary endpoint is the frequency of DLTs which are relevant for the determination the tentative RP2D in Part 1 of the trial.
Part 2, Cohort 2 (phase IIa - melanoma): Disease control (DC) according to RECIST 1.1 | up to 12 weeks from treatment start
  DC is defined as any complete response (CR), partial response (PR) or stable disease (SD) for 12 weeks from start of treatment according to RECIST 1.1 criteria achieved during trial treatment. Any patient with CR, PR or SD (≥ 12 weeks) as best observed response during trial treatment will be considered as a success; otherwise they will be considered as a failure.
  Patients without any response assessment during trial treatment will be regarded as having a non-evaluable response (NE) and thus will be considered as failures for this endpoint.

SECONDARY OUTCOMES:
Objective response according to iRECIST (iOR) | up to 12 weeks from treatment start
  iOR is defined as any complete response (CR/iCR) or partial response (PR/iPR) according to RECIST 1.1 or iRECIST criteria achieved during trial treatment until disease progression according to iRECIST, death or subsequent anticancer treatment, whichever occurs first. Any patient with CR/iCR or PR/iPR as best observed response during trial treatment until disease progression according to iRECIST, death or subsequent anticancer treatment (whichever occurs first) will be considered as a success; otherwise they will be considered as a failure.
  Patients without any objective response assessment during trial treatment until disease progression according to iRECIST, death or subsequent anticancer treatment (whichever occurs first) will be regarded as having a NE and thus will be considered as failures for this endpoint.
Disease control according to iRECIST (iDC) | up to 12 weeks from treatment start
  iDC is defined as any complete response (CR/iCR), partial response (PR/iPR) or stable disease (SD/iSD) for 12 weeks according to RECIST 1.1 or iRECIST criteria achieved during trial treatment until disease progression according to iRECIST, death or start of a subsequent anticancer treatment, whichever occurs first. Any patient with CR/iCR, PR/iPR or SD/iSD (≥12 weeks) as best observed response during trial treatment until disease progression according to iRECIST, death or start of a subsequent anticancer treatment (whichever occurs first) will be considered as a success; otherwise they will be considered as a failure.
  Patients without any response assessment during trial treatment until disease progression according to iRECIST, death or start of a subsequent anticancer treatment (whichever occurs first) will be regarded as having a NE and thus will be considered as failures for this endpoint.
Duration of response according to iRECIST (iDoR) | from date of response until date of disease progression according to iRECIST or death due to disease progression, whichever occurs first, assessed up to 4 years
  iDoR is defined as the time from the first documentation of iOR until disease progression according to iRECIST criteria (iPD) or death due to disease progression.
  iPD is defined as the time point of first iUPD without subsequent iSD, iPR or iCR before trial treatment discontinuation.
  Patients not experiencing an event at the time of the analysis, as well as patients starting a subsequent anticancer treatment in the absence of an event, will be censored at the date of their last available tumor assessment showing no evidence of iPD before starting a subsequent anticancer treatment, if any.
Progression-free survival according to iRECIST (iPFS) | from treatment start until date of disease progression according to iRECIST or death due to any reason, whichever occurs first, assessed up to 4 years
  iPFS is defined as the time from treatment start until disease progression according to iRECIST criteria (iPD) or death due to any reason, whichever occurs first.
  iPD is defined as the time point of first iUPD without subsequent iSD, iPR or iCR before trial treatment discontinuation.
  Patients not experiencing an event at the time of the analysis, as well as patients starting a subsequent anticancer treatment in the absence of an event, will be censored at the date of their last available tumor assessment before starting a subsequent anticancer treatment, if any.
Objective response (OR) according to RECIST 1.1 | up to 24 weeks from treatment start
  OR is defined as any complete response (CR) or partial response (PR) according to RECIST 1.1 criteria achieved during trial treatment. Any patient with CR or PR as best observed response during trial treatment will be considered as a success; otherwise they will be considered as a failure.
  Patients without any objective response assessment during trial treatment will be regarded as having a NE and thus will be considered as failures for this endpoint.
Disease control (DC) according to RECIST 1.1 (only for Part 2, Cohort 1) | up to 24 weeks from treatment start
  DC is defined as any complete response (CR), partial response (PR) or stable disease (SD) for 12 weeks from registration according to RECIST 1.1 criteria achieved during trial treatment. Any patient with CR, PR or SD (≥ 12 weeks) as best observed response during trial treatment will be considered as a success; otherwise they will be considered as a failure.
  Patients without any response assessment during trial treatment will be regarded as having a NE and thus will be considered as failures for this endpoint.
Duration of response (DoR) according to RECIST 1.1 | from date of response until date of disease progression according to RECIST 1.1 or death due to disease progression, whichever occurs first, assessed up to 4 years
  DoR is defined as the time from the first documentation of OR until disease progression according to RECIST 1.1 criteria or death due to disease progression, whichever occurs first.
  Patients not experiencing an event at the time of the analysis, as well as patients starting a subsequent anticancer treatment in the absence of an event, will be censored at the date of their last available tumor assessment before starting a subsequent anticancer treatment, if any.
Progression-free survival (PFS) according to RECIST 1.1 | from treatment start until date of disease progression according to RECIST 1.1 or death due to any reason, whichever occurs first, assessed up to 4 years
  PFS is defined as the time from treatment start until disease progression according to RECIST 1.1 criteria or death due to any reason, whichever occurs first.
  Patients not experiencing an event at the time of the analysis, as well as patients starting a subsequent anticancer treatment in the absence of an event, will be censored at the date of their last available tumor assessment before starting a subsequent anticancer treatment, if any.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Joerger, MD PhD, Study Chair — Cantonal Hospital of St. Gallen
Locations (3):
- Switzerland (3):
  - Inselspital, Bern, Bern
  - Kantonsspital Graubünden, Chur
  - Kantonsspital St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No